CLINICAL TRIAL: NCT05010850
Title: SafeHeal Colovac Colorectal Anastomosis Protection Device Evaluation (SAFE-2) Pivotal Study: A Study to Evaluate the Safety and Effectiveness of the Colovac Colorectal Anastomosis Protection Device
Brief Title: SafeHeal Colovac Colorectal Anastomosis Protection Device Evaluation (SAFE-2) Pivotal Study
Acronym: SAFE-2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Voluntary and temporary suspension of enrollment.
Sponsor: SafeHeal Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAFE-2
Record Dates: First submitted 2021-08-11; First posted 2021-08-18 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer; Rectal Cancer; Rectal Tumor; Rectal/Anal
Keywords: anastomosis; leak; colorectal; ileostomy
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Colovac (Experimental): Patients receive Colovac during colorectal surgery
  Interventions: Device: Colovac
- Standard of Care (Active Comparator): Patients receive the standard of care, a protective stoma, during colorectal surgery
  Interventions: Procedure: Stoma Creation

INTERVENTIONS:
Device: Colovac — A removable, temporary intraluminal bypass device designed to safely postpone the creation of a protective stoma until 10 days after surgery for only patients who need it (do not have a healed anastomosis)
  Arms: Colovac
Procedure: Stoma Creation — Protective ileostomy
  Arms: Standard of Care

SUMMARY:
A randomized trial to assess the safety and effectiveness of the Colovac in providing temporary protection of the anastomosis in subjects undergoing lower anterior resection for colorectal cancer.

DETAILED DESCRIPTION:
A primary diverting stoma is widely used by surgeons in order to bypass the low rectal anastomosis and reduce morbidity associated with anastomotic leaks. Typically, a stoma is created for all high-risk patients which means that many patients are exposed to potentially serious complications associated with the stoma itself without any clinical benefit.

Colovac is a local, temporary, minimally invasive bypass device that provides protection of the anastomosis and safely postpones stoma creation for 10 days after surgery. By postponing stoma creation for 10 days, Colovac is designed to avoid stoma creation in all patients except those patients whose anastomoses have not healed by 10 days after surgery, allowing the others to return to normal activity more quickly and safely.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (greater than 18 years of age)
2. Eligible to undergo open or minimally invasive sphincter-preserving lower anterior resection (anastomosis within 10 cm of the anal verge) with planned diverting loop ileostomy for malignant indication, assessed by a multi-disciplinary team.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2
4. Willing to comply with protocol-specific treatment and study visits and to sign a written Informed Consent Form

Exclusion Criteria:

1. History of left colitis
2. Known allergy to nickel or other components of the Colovac kit
3. Pregnant or nursing female subject
4. Concomitant major surgical procedure in combination with Colorectal resection (e.g.. hepatectomy)
5. Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation, impair the ability of the participant to undergo protocol described procedures or interfere with the interpretation of study results. including, but not limited to:

   1. COVID-19 positive (active infection) if test required by hospital
   2. Immunodeficiency (CD4+ count < 500 mm3)
   3. Systemic steroid therapy within the past 6 months
   4. Systemic infection at the time of surgery or requiring systemic antimicrobial therapy up to 1 week before surgery
   5. Major surgical or interventional procedures within 30 days prior to this study or planned surgical or interventional procedures within 30 days of entry into this study
   6. Diagnosis of bowel obstruction, bowel strangulation, peritonitis, bowel perforation, intraabdominal infection, ischemic bowel, carcinomatosis
   7. Fecal incontinence, involvement of sphincter by the neoplastic disease or evidence of extensive local disease in the pelvis seen on pre-operative imaging
   8. Severe Malnutrition defined as ≥ 10% weight loss within 3 months prior to enrollment
   9. Stage IV colorectal cancer unless curative intent R0 resection is planned AND there is no associated peritoneal disease
6. The subject is currently participating in another investigational drug or device study
7. Occurrence of any of the following during the colorectal surgery:

   1. Blood loss (>750 cc)
   2. Blood transfusion
   3. Any new sign of ischemia
   4. Positive air leak test
   5. Inadequate bowel preparation
   6. Anastomosis location greater than 10 cm from the anal verge
   7. Other intra-operative risks that preclude the subject from undergoing the procedure with the investigational device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Sylla, MD, Principal Investigator — MOUNT SINAI HOSPITAL; Jeremie Lefevre, MD, PhD, Principal Investigator — Hopital Saint Antoine
Locations (16):
- United States (10):
  - Kaiser Permanente - Los Angeles, Los Angeles, California
  - USC Keck Hospital, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Tampa General Hospital, Tampa, Florida
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Dartmouth-Hitchcock, Lebanon, New Hampshire
  - Maimonides Medical Center, Brooklyn, New York
  - Mount Sinai Hospital, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Lankenau Medical Center, Wynnewood, Pennsylvania
- Universitair Ziekenhuis Antwerpen, Edegem, Antwerp, Belgium
- France (5):
  - CHU de Besancon, Besançon
  - ICM Val d'Aurelle, Montpellier
  - Hopital Saint-Louis, Paris
  - CHU Rouen Normandie, Rouen
  - Hôpital Saint Antoine Paris, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hain E, Lefevre JH, Ricardo A, Lee S, Zaghiyan K, McLemore E, Sherwinter D, Rhee R, Wilson M, Martz J, Maykel J, Marks J, Marcet J, Rouanet P, Maggiori L, Komen N, De Hous N, Lakkis Z, Tuech JJ, Attiyeh F, Cotte E, Sylla P. SafeHeal Colovac Colorectal Anastomosis Protection Device evaluation (SAFE-2) pivotal study: an international randomized controlled study to evaluate the safety and effectiveness of the Colovac Colorectal Anastomosis Protection Device. Colorectal Dis. 2024 Jun;26(6):1271-1284. doi: 10.1111/codi.17012. Epub 2024 May 15. PMID 38750621

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Following intra-operative exclusion apply which may have prevented subjects from being enrolled after signing consent: Occurrence of any of the following during colorectal surgery:
  1. Blood loss (>750 cc)
  2. Blood transfusion
  3. Any new sign of ischemia
  4. Positive air leak test
  5. Inadequate bowel preparation
  6. Anastomosis location greater than 10 cm from the anal verge
  7. Other intra-operative risks that preclude the subject from undergoing the procedure with the investigational device
Period: Overall Study
Arm/Group | Colovac | Standard of Care
Started | 10 | 8
Completed | 8 | 6
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Colovac | Standard of Care | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] — Age of subjects which were enrolled and analyzed in the study
  years | 67.1 (10.9) | 60.9 (11.4) | 64.3 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Percentages Female and Male
  Participants
    Female | 6 | 3 | 9
    Male | 4 | 5 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Mean Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 24.8 (5.5) | 25.7 (4.8) | 25.2 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Avoidance of Ostomy
Description: Reduction in stoma creation rate
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Colovac | Standard of Care
Number analyzed (Participants) | 10 | 8
Participants | 7 | 0

2. Primary Outcome: Safety Major Complications
Description: Rate of subjects with major complications
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Colovac | Standard of Care
Number analyzed (Participants) | 10 | 8
Participants | 3 | 2

ADVERSE EVENTS:
Time Frame: 1 year
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Standard of Care | Colovac
All-Cause Mortality (participants affected / at risk) | 1/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 7/8 | 6/10
Other Adverse Events (participants affected / at risk) | 6/8 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=8) | Colovac (N=10)
General state of deterioration with dehydration, resulting in death (General disorders) | 1 (1) | 0 (0) — not related to the Low Anterior Resection Surgery or the stoma
Anastomosis Leakage (General disorders) | 2 (2) | 4 (4) — Causally related to the Low Anterior Resection surgery
Undernutrition with Naso Gastric Tube (Gastrointestinal disorders) | 1 (1) | 0 (0) — Probably or causally related to the stoma
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) — Probably or causally related to the stoma
Colon Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1) — Causally related to the Colovac device
Acute Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1) — Probably related to the stoma reversal procedure
Infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
CRP Elevation (Infections and infestations) | 1 (1) | 0 (0)
Dehydration which resolved (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=8) | Colovac (N=10)
Abdominal/ Anal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anastomosis leakage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholestasis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haematuria (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Heart Failure (Cardiac disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Incisional hernia (Surgical and medical procedures) | 0 (0) | 1 (1)
Infection of incision/surgery wound on left side (Surgical and medical procedures) | 1 (1) | 0 (0)
Inflammation of skin around the anus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea/vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nerve Tissue Injury (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Other - Denutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Other - Epigastric Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Other - Lymphopenia to Xeloda (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Other - Polyneuropathie (Nervous system disorders) | 1 (1) | 1 (1)
Other - Renal Failure (Endocrine disorders) | 1 (1) | 0 (0)
Other - Worsening Hernia Inguinalis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Parastomal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary Infection (Endocrine disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The SAFE-2 study was voluntarily terminated early by the sponsor due to non-safety reasons. Given the limited sample size of SAFE-2, further studies with larger cohorts are recommended.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/50/NCT05010850/Prot_SAP_001.pdf